CLINICAL TRIAL: NCT06977139
Title: Interventional Structural Registry - LuEbeck
Acronym: INSTYLE
Status: Recruiting | Type: Observational
Sponsor: Prof. Dr. med. Ingo Eitel (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Ingo Eitel, Head of Department, University of Luebeck
Organization: University of Luebeck (Other)
Other Study IDs: 21-330; 21-330 (Registry Identifier: INSTYLE)
Record Dates: First submitted 2025-05-08; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Structural Heart Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the registry is to investigate the effect of catheter-assisted procedures in the context of structural heart disease on clinical morbidity and mortality. Furthermore, the long-term prognosis of patients after a catheter-based procedure is to be evaluated.

In particular, the following parameters will be documented and the following questions discussed:

* Underlying and concomitant diseases of these patients
* Evaluation of the methods in relation to the respective disease
* Safety - acute and long-term
* Effectiveness - periprocedural, hospital and long-term course
* Concomitant therapies

ELIGIBILITY:
Inclusion Criteria:

* Structural heart disease

Exclusion Criteria:

* Patients without consent/information
* Age ≤ 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients for who the indication for a catheter-based heart valve replacement or closure system was set due to a structural heart disease can be included.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-09-11 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Combined endpoint | 30days
  Combined endpoint of NYHA classification, re-hospitalization, death, repeat procedure, heart transplantation, LVAD implantation (the order is not relevant) by day 30.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: Undecided